CLINICAL TRIAL: NCT01941836
Title: A Randomized, Double-Blind, Parallel Group, Multicenter Study to Evaluate the Efficacy and Safety of ETC-1002, Ezetimibe, and the Combination in Hypercholesterolemic Patients With or Without Statin Intolerance
Brief Title: Evaluation of ETC-1002, Ezetimibe, and the Combination in Hypercholesterolemic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Esperion Therapeutics, Inc. (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1002-008
Record Dates: First submitted 2013-09-06; First posted 2013-09-13 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Hypercholesterolemia
Keywords: Statin intolerant; Statin tolerant; LDL; Cholesterol
MeSH Terms: conditions — Hypercholesterolemia | interventions — 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid; Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- ETC-1002 120 mg/day (Experimental): Orally, once daily in morning as capsules
  Interventions: Drug: ETC-1002
- ETC-1002 180 mg/day (Experimental): Orally, once daily in morning as capsules
  Interventions: Drug: ETC-1002
- ezetimibe 10mg/day (Active Comparator): Orally, once daily in morning as capsules
  Interventions: Drug: Ezetimibe
- ETC-1002 120 mg/day + ezetimibe 10mg/day (Experimental): Orally, once daily in morning
  Interventions: Drug: ETC-1002; Drug: Ezetimibe
- ETC-1002 180 mg/day + ezetimibe 10mg/day (Experimental): Orally, once daily in morning
  Interventions: Drug: ETC-1002; Drug: Ezetimibe

INTERVENTIONS:
Drug: ETC-1002 — Patients receive ETC-1002
  Arms: ETC-1002 120 mg/day; ETC-1002 120 mg/day + ezetimibe 10mg/day; ETC-1002 180 mg/day; ETC-1002 180 mg/day + ezetimibe 10mg/day
Drug: Ezetimibe — Patients receive ezetimibe
  Other Names: Zetia
  Arms: ETC-1002 120 mg/day + ezetimibe 10mg/day; ETC-1002 180 mg/day + ezetimibe 10mg/day; ezetimibe 10mg/day

SUMMARY:
The purpose of this research study is to see how ETC-1002 is tolerated in the body, to measure the amount of ETC-1002 in the blood, and to determine how ETC-1002 affects the level of LDL-cholesterol (bad cholesterol) and other markers of health and disease in blood and urine in patients with elevated LDL-cholesterol with or without statin intolerance.

DETAILED DESCRIPTION:
Hypercholesterolemic patients either with or without a history of statin intolerance (1:1 ratio) will be randomized to receive once daily by mouth capsules containing either ETC-1002, ezetimibe, or ETC-1002 + ezetimibe. This study will explore the safety and efficacy of concomitant administration of ETC-1002 and ezetimibe, while also exploring the effect of ezetimibe on ETC-1002 systemic exposure.

ELIGIBILITY:
Key Inclusion Criteria:

* Statin intolerant and statin tolerant
* Fasting LDL-C between 130 mg/dL and 220 mg/dL
* Fasting triglyceride less than or equal to 400 mg/dL
* Body mass index (BMI) between 18 and 45 kg/m2

Key Exclusion Criteria:

* History or current clinically significant cardiovascular disease
* History or current type 1 diabetes or uncontrolled type 2 diabetes
* Use of metformin or thiazolidinediones (TZD) within 3 months of screening
* History of joint symptoms difficult to differentiate from myalgia
* Uncontrolled hypothyroidism
* Liver disease or dysfunction
* Renal dysfunction or nephritic syndrome
* Gastrointestinal (GI) conditions or prior GI procedures
* HIV or AIDS
* History or malignancy
* History or drug or alcohol abuse within last 2 years
* Use of experimental or investigational drugs within 30 days of screening
* Use of ETC-1002 in a previous clinical study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2013-09; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Percent change in calculated low density lipoprotein-cholesterol (LDL-C) | Baseline and 12 weeks

SECONDARY OUTCOMES:
Percent change in other lipid measures non high density lipoprotein cholesterol (nonHDL-C) | Baseline and 12 weeks
Safety using adverse event reports; vital signs | up to 21 weeks including screening
Percent change in Apolipoprotein B (ApoB) | Baseline and 12 weeks
Percent change in high sensitivity C-reactive protein (hsCRP) | Baseline and 12 weeks
Safety using adverse event reports; clinical laboratory results | up to 21 weeks including screening
Safety using adverse event reports; rates of muscle-related adverse | up to 21 weeks including screening

OTHER OUTCOMES:
Pharmacokinetic plasma trough concentrations of ETC-1002 and its metabolite ESP15228 | Week 2, Week 4, Week 8 and Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Diane E MacDougall, MS, Study Director — Esperion Therapeutics, Inc.
Locations (64):
- United States (64):
  - Birmingham, Alabama
  - Muscle Shoals, Alabama
  - Chandler, Arizona
  - Beverly Hills, California
  - Chino, California
  - Lincoln, California
  - Long Beach, California
  - Los Angeles, California
  - Newport Beach, California
  - Thousand Oaks, California
  - Vista, California
  - Denver, Colorado
  - Hartford, Connecticut
  - Atlantis, Florida
  - Brandon, Florida
  - Hialeah, Florida
  - Jacksonville, Florida
  - Oviedo, Florida
  - Ponte Vedra, Florida
  - Port Orange, Florida
  - St. Petersburg, Florida
  - West Palm Beach, Florida
  - Decatur, Georgia
  - Marietta, Georgia
  - Meridian, Idaho
  - Evansville, Indiana
  - Kansas City, Kansas
  - Auburn, Maine
  - Lincoln, Nebraska
  - Clifton, New Jersey
  - Albuquerque, New Mexico
  - New Windsor, New York
  - Rochester, New York
  - Williamsville, New York
  - Greensboro, North Carolina
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Wilmington, North Carolina
  - Beachwood, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Franklin, Ohio
  - Lyndhurst, Ohio
  - Marion, Ohio
  - Willoughby Hills, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Eugene, Oregon
  - Mt. Pleasant, South Carolina
  - Kingsport, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Round Rock, Texas
  - Orem, Utah
  - Salt Lake City, Utah
  - Norfolk, Virginia
  - Richmond, Virginia
  - Olympia, Washington
  - Renton, Washington
  - Seattle, Washington
  - Spokane, Washington

REFERENCES:
- [Background] Ballantyne CM, Davidson MH, Macdougall DE, Bays HE, Dicarlo LA, Rosenberg NL, Margulies J, Newton RS. Efficacy and safety of a novel dual modulator of adenosine triphosphate-citrate lyase and adenosine monophosphate-activated protein kinase in patients with hypercholesterolemia: results of a multicenter, randomized, double-blind, placebo-controlled, parallel-group trial. J Am Coll Cardiol. 2013 Sep 24;62(13):1154-62. doi: 10.1016/j.jacc.2013.05.050. Epub 2013 Jun 13. PMID 23770179
- [Background] Filippov S, Pinkosky SL, Lister RJ, Pawloski C, Hanselman JC, Cramer CT, Srivastava RAK, Hurley TR, Bradshaw CD, Spahr MA, Newton RS. ETC-1002 regulates immune response, leukocyte homing, and adipose tissue inflammation via LKB1-dependent activation of macrophage AMPK. J Lipid Res. 2013 Aug;54(8):2095-2108. doi: 10.1194/jlr.M035212. Epub 2013 May 24. PMID 23709692
- [Background] Pinkosky SL, Filippov S, Srivastava RA, Hanselman JC, Bradshaw CD, Hurley TR, Cramer CT, Spahr MA, Brant AF, Houghton JL, Baker C, Naples M, Adeli K, Newton RS. AMP-activated protein kinase and ATP-citrate lyase are two distinct molecular targets for ETC-1002, a novel small molecule regulator of lipid and carbohydrate metabolism. J Lipid Res. 2013 Jan;54(1):134-51. doi: 10.1194/jlr.M030528. Epub 2012 Nov 1. PMID 23118444
- [Background] Gutierrez MJ, Rosenberg NL, Macdougall DE, Hanselman JC, Margulies JR, Strange P, Milad MA, McBride SJ, Newton RS. Efficacy and safety of ETC-1002, a novel investigational low-density lipoprotein-cholesterol-lowering therapy for the treatment of patients with hypercholesterolemia and type 2 diabetes mellitus. Arterioscler Thromb Vasc Biol. 2014 Mar;34(3):676-83. doi: 10.1161/ATVBAHA.113.302677. Epub 2014 Jan 2. PMID 24385236
- [Derived] Thompson PD, MacDougall DE, Newton RS, Margulies JR, Hanselman JC, Orloff DG, McKenney JM, Ballantyne CM. Treatment with ETC-1002 alone and in combination with ezetimibe lowers LDL cholesterol in hypercholesterolemic patients with or without statin intolerance. J Clin Lipidol. 2016 May-Jun;10(3):556-67. doi: 10.1016/j.jacl.2015.12.025. Epub 2016 Jan 6. PMID 27206943